CLINICAL TRIAL: NCT05343689
Title: Effect of the Pneumatic Compression of Lower Leg on Post-induction Hypotension in Elderly Patients Undergoing Robot Assisted Laparoscopic Prostatectomy: a Double Blined Randomized Controlled Trial
Brief Title: Pneumatic Compression and Post-induction Hypotension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, MD, Principal Investigator, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-0495
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pneumatic compression group (Experimental): When inducing general anesthesia, pneumatic compression is performed.
  Interventions: Procedure: Pneumatic compression
- Control group (No Intervention): When inducing general anesthesia, pneumatic compression is not performed.

INTERVENTIONS:
Procedure: Pneumatic compression — Pneumatic compression with preset pressure and cyclic manner is applied from immediately after anesthesia induction to 20 minutes after anesthesia induction in the both legs.
  Arms: Pneumatic compression group

SUMMARY:
The purpose of this study is to evaluate the effect of pneumatic compression on post-induction hypotension in elderly patients undergoing robot assisted laparoscopic prostatectomy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of pneumatic compression of lower leg, which is performed during 20 minutes after anesthesia induction period, on post-induction hypotension in elderly patients undergoing robot assisted laparoscopic prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled robot assisted laparoscopic prostatectomy under general anesthesia
* Elderly patients (between 65 and 79 years old)
* American Society of Anesthesiologists physical status ≤3
* Patients who are voluntarily agreed to this clinical study

Exclusion Criteria:

* Uncontrolled hypertension, heart failure (ejection fraction <40%), arrhythmia requiring treatment, unstable coronary artery disease
* Patient's denial

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

PRIMARY OUTCOMES:
Incidence of post-induction hypotension | From anesthesia induction to 20 minutes after anesthesia induction
  Systolic blood pressure below 90 mmHg

SECONDARY OUTCOMES:
Blood pressure | From anesthesia induction to 20 minutes after anesthesia induction
  Blood pressure (systolic, diastolic, and mean)
Heart rate | From anesthesia induction to 20 minutes after anesthesia induction
  Heart rate derived from electrocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reich DL, Hossain S, Krol M, Baez B, Patel P, Bernstein A, Bodian CA. Predictors of hypotension after induction of general anesthesia. Anesth Analg. 2005 Sep;101(3):622-628. doi: 10.1213/01.ANE.0000175214.38450.91. PMID 16115962
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Geerts WH, Bergqvist D, Pineo GF, Heit JA, Samama CM, Lassen MR, Colwell CW. Prevention of venous thromboembolism: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines (8th Edition). Chest. 2008 Jun;133(6 Suppl):381S-453S. doi: 10.1378/chest.08-0656. PMID 18574271
- [Background] Golparvar M, Saghaei M, Saadati MA, Farsaei S. Effect of ondansetron on prevention of post-induction hypotension in elderly patients undergoing general anesthesia: A randomized, double-blind placebo-controlled clinical trial. Saudi J Anaesth. 2015 Oct-Dec;9(4):365-9. doi: 10.4103/1658-354X.159455. PMID 26543450